CLINICAL TRIAL: NCT05682547
Title: A Single Center, Randomized, Controlled Trial Comparing the Clinical Efficacy of 3% Diquafosol Tetrasodium and 0.1 % Hyaluronic Acid 0.1% in Diabetic Patients With Dry Eye Disease
Brief Title: Diquafosol vs Hyaluronic Acid for Diabetic Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: He Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DMDEDQS-2022-12
Record Dates: First submitted 2022-12-05; First posted 2023-01-12 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2024-05

CONDITIONS: Diabetic Eye Problems
Keywords: Dry eye; Diquafosol; Hyaluronate; Diabetic dry eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Lubricant Eye Drops

STUDY DESIGN:
Intervention Model Description: Prospective, randomised control trial.
Who Masked: Outcomes Assessor
Masking Description: Masked examiner for all clinical assessments will not involved in the data collection or group allocation procedure for this research. The investigator will not be aware of the two groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DQS group (Experimental): Participants in DQS group will be administered one drop of 3% DQS (Diquas, Santen Pharmaceutical Co., Ltd., Osaka, Japan) six times per day for 8 weeks.
  Interventions: Drug: 3% Diquafosol tetrasodium
- HA group (Active Comparator): Participants in HA group will be administered one drop of 0.1% Sodium hyaluronate artificial tears (preservative free) six times per day for 8 weeks
  Interventions: Drug: 0.1% hyaluronate

INTERVENTIONS:
Drug: 3% Diquafosol tetrasodium — 3% Diquafosol tetrasodium eye drops will be used to assess its usefulness in diabetic dry eye symptoms
  Other Names: Diquas
  Arms: DQS group
Drug: 0.1% hyaluronate — 0.1% hyaluronate eye drops will be used to assess its usefulness in diabetic dry eye symptoms and compared to 3% Diquafosol tetrasodium eye drops.
  Other Names: Artificial tears
  Arms: HA group

SUMMARY:
Diquafosol ophthalmic solution (DQS) stimulates P2Y2 receptors on the ocular surface, which enhances mucin secretion from goblet cells. Therefore, tear film stability and hydration of the ocular surface can be achieved independent from lacrimal glands function. While it has been observed that 0.1 percent hyaluronate (HA) in artificial tears promotes corneal re-epithelium and improves corneal healing.This prospective, open label pilot study will include 60 eyes of 30 diabetic patients diagnosed with DED and will be randomly assigned to either DQS (n=30 eyes) or ATD group (n=30 eyes). Participants in the DQS group will receive 3% Diquafosol ophthalmic solution, while HA group will receive 0.1% Sodium hyaluronate artificial tears. The dosage for both drugs will be one drop, six times per day for 4 weeks. Tear film lipid layer (TFLL), non-invasive breakup time (NITBUT), corneoconjunctival staining score (CS), meibum gland (MG), conjunctival hyperemia (RS score), ocular surface disease index (OSDI) will be assessed and compared at baseline, day-14, and day-28.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is a prevalent chronic metabolic illness that causes relative insulin insufficiency in target organs owing to pancreatic β-cell dysfunction and insulin resistance [1]. Shift to sedentary lifestyle, ageing population and obesity has significantly contributed to the global rise in the prevalence of T2DM [2]. In 2019 the prevalence of diabetes was documented to be 9.3% (463 million people) and in 2030 it is estimated to rise to 10.2% (578 million) and T2DM accounts for approximately 90% of all diabetic occurrence[3]. Negative alterations to the tear film, corneal epithelium, corneal endothelium, and corneal nerves have been observed in 47-64% of patients with diabetes[4] [5]. Ocular surface manifestation of signs and symptoms secondary to DM has been termed as diabetic keratopathy (DK). DK has been documented to increase central corneal thickness[6], decrease in endothelial cell density[7], leads of superficial punctate keratitis[8], delay and impede wound repair[9], and decrease in corneal sensitivity due to neuropathy[10]. Additionally, DM patients have also been noted to have compromised tear quantity and quality[11][12] due to conjunctival goblet cell loss as documented on cytologic analysis [13]. Goblet cells secrete mucin, which stabilizes the tear film, minimizes tear evaporation, and reduces mechanical friction. Goblet cell loss in animal models suggests that it disrupts the ocular surface's immune tolerance [14] and increased expression of inflammatory cytokines in the conjunctiva[15]. 0.1% hyaluronate (HA) used in artificial tears have been reported to promote corneal re-epithelium and improve corneal healing[16].

Additionally, HA has been reported to decrease the rate of tear evaporation and enhance the stability of tear film [17]. Diquafosol tetrasodium is a dinucleotide polyphosphate which a purinoceptor agonist, when administered to the ocular surface, it binds to P2Y2 receptors and stimulates mucin and tear secretion[18-20]. The corneal epithelium, conjunctival epithelium, lacrimal gland ductal epithelium, meibomian gland sebaceous cells, and meibomian gland ductal cells all express the P2Y2 receptor. [21,22]. Subsequently, enhanced secretion of mucin and tear secretion due to Diquafosol tetrasodium ophthalmic solution (DQS) stabilize the tear film, minimizes tear evaporation, and reduces mechanical friction thereby protecting the corneal epithelium [23]. Various reports have concluded that that 3% DQS is effective in the treatment of dry eye disease [24-26] and Current [19] findings suggest that DQS improves corneal epithelial damage in T2DM rat model.

However, the effect of DQS on the tear film of T2DM humans has not been previously assessed. Therefore, the purpose s to assess subjective and objective diabetic dry eye findings after using 3% DQS or 0.1% HA topical eye drops.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Clinical diagnosed and confirmed with type 2 diabetes for one year or more
* Able and willing to comply with the treatment/follow-up schedule
* Bilateral signs and symptoms of dry eye disease

Exclusion Criteria:

* Participants with systemic immune-mediated illnesses, such as secondary Sjögren's syndrome or graft-versus-host disease
* Patients using topical medication(s) for the treatment of ocular disorders such as glaucoma or allergic conjunctivitis were excluded from the study.
* Previous ocular surgery or trauma
* 1-month history of blepharal and periorbital skin disease or allergies
* Severe dry eyes with corneal epithelial defect
* Limbic keratitis
* Pterygium
* Corneal neovascularization
* Glaucoma
* Breastfeeding
* Rheumatic immune systemic diseases
* Herpes zoster infection
* Pregnant women
* Allergic to fluorescein
* Contact lens wearers

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Non-invasive tear break-up time | Day-0 (baseline), week-4, and week-8
  Non-invasive initial tear film breaking time will be assessed using the Keratograph 5M (Oculus, Germany) topographer. Three sequentially readings will be captured, and the median value will be included in the final analysis. The median value will be recorded.
  * Changes at week-4, and week-8 will be compare with baseline measurements.
  * Comparison between groups at baseline, week-4, and week-8 will also be examined.

SECONDARY OUTCOMES:
Conjunctival hyperemia (RS score) | Day-0 (baseline), week-4, and week-8
  Conjunctival hyperemia (RS score) will be assessed by keratograph image (Oculus, Germany) of 1156*873 pixels, redness score (RS) (accurate to 0.1 U) was displayed on the computer screen that ranged from 0.0 to 4.0.
  * Changes at week-4, and week-8 will be compare with baseline measurements.
  * Comparison between groups at baseline, week-4, and week-8 will also be examined.
Quality of meibum grade | Day-0 (baseline), week-4, and week-8
  Meibum quality will be assessed under a slit-lamp:
  Five meibomian gland in the middle parts of the eyelid will be assessed using a scale of 0 to 3 for each gland (0 represented clear meibum; 1 represented cloudy meibum; 2 represented cloudy and granular meibum; and 3 represented thick, toothpaste like consistency meibum).
  * Changes at week-4, and week-8 will be compare with baseline measurements.
  * Comparison between groups at week-4, and week-8 will also be examined.
Expressibility of meibum grade | Day-0 (baseline), week-4, and week-8
  Meibum expressibility will be assessed under a slit-lamp:
  Eight meibomian glands in the middle part will be evaluated on a scale of 0 to 3 (0 denoted that all glands expressible; 1 denoted that 3 to 4 glands expressible; 2 denoted those 1 to 2 glands expressible; and 3 denoted that no glands were expressible). The overall score was computed using the mean scores of these eight glands.
  * Changes at week-4, and week-8 will be compare with baseline measurements.
  * Comparison between groups at baseline, week-4, and week-8 will also be examined.
Conjunctivocorneal epithelial staining grade | Day-0 (baseline), week-4, and week-8
  Conjunctivocorneal epithelial staining will be assessed under a slit-lamp:
  Conjunctivocorneal epithelial staining will be assess corneal and conjunctival epithelium damage. Double vital staining approach with two microliters of a preservative-free solution containing 1% lissamine green and 1% sodium fluorescein will be instilled in the conjunctival sac.
  The eye will be sectioned into three equal pieces (temporal conjunctiva, cornea, and nasal conjunctiva). Each region receives a maximum staining score of three points and a minimum of zero points. The combined scores from all three parts were then recorded on a scale ranging from 0 (normal) to 9 (severe).
  * Changes at week-4, and week-8 will be compare with baseline measurements.
  * Comparison between groups at baseline, week-4, and week-8 will also be examined.
Tear Film Lipid Layer | Day-0 (baseline), week-4, and week-8
  Tear Film Lipid Layer interferometry will be assessed using DR-1 (Kowa, Nagoya, Japan).
  * Changes at week-4, and week-8 will be compare with baseline measurements.
  * Comparison between groups at baseline, week-4, and week-8 will also be examined.
OSDI Score | Day-0 (baseline), week-4, and week-8
  Chinese translated, and validated OSDI (Allergan Inc, Irvine, USA) version will beused to assess and quantify DE symptom. The 12 items of the questionnaire can be tabulated into a score that ranges from 0 (no symptoms) to 100 (severe symptoms) points
  * Changes at week-4, and week-8 will be compare with baseline measurements.
  * Comparison between groups at baseline, week-4, and week-8 will also be examined.
Tear meniscus height (TMH) | Day-0 (baseline), week-4, and week-8
  Tear meniscus height using the Keratograph 5M (Oculus, Germany) topographer
Corneal Sensitivity Score | Day-0 (baseline), week-4, and week-8
  Corneal Sensitivity Score measured with Cochet-Bonnet esthesiometer (in mm filament length)
Corneal nerves and immune/inflammatory cells change | Day-0 (baseline), week-4, and week-8
  HRT III RCM, (Heidelberg Engineering GmbH, Dossenheim, Germany) will be used to record corneal nerves and immune/inflammatory cells change.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Eric Pazo, Study Chair — He Eye Hospital, Shenyang, China
Locations (1):
- He Eye Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes
The study's findings will be shared regardless of the effect's direction. All possible beneficiaries of the research, including patients, carers, family, doctors, advisory boards, and medical boards, will receive trial data. Publications in high-impact, open-access medical journals and talks at national and international medical conferences will serve this purpose.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Result] Chatterjee S, Khunti K, Davies MJ. Type 2 diabetes. Lancet. 2017 Jun 3;389(10085):2239-2251. doi: 10.1016/S0140-6736(17)30058-2. Epub 2017 Feb 10. PMID 28190580
- [Result] Weisman A, Fazli GS, Johns A, Booth GL. Evolving Trends in the Epidemiology, Risk Factors, and Prevention of Type 2 Diabetes: A Review. Can J Cardiol. 2018 May;34(5):552-564. doi: 10.1016/j.cjca.2018.03.002. Epub 2018 Mar 13. PMID 29731019
- [Result] Saeedi P, Petersohn I, Salpea P, Malanda B, Karuranga S, Unwin N, Colagiuri S, Guariguata L, Motala AA, Ogurtsova K, Shaw JE, Bright D, Williams R; IDF Diabetes Atlas Committee. Global and regional diabetes prevalence estimates for 2019 and projections for 2030 and 2045: Results from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2019 Nov;157:107843. doi: 10.1016/j.diabres.2019.107843. Epub 2019 Sep 10. PMID 31518657
- [Result] Abdelkader H, Patel DV, McGhee CNj, Alany RG. New therapeutic approaches in the treatment of diabetic keratopathy: a review. Clin Exp Ophthalmol. 2011 Apr;39(3):259-70. doi: 10.1111/j.1442-9071.2010.02435.x. Epub 2011 Apr 4. PMID 20973888
- [Result] Vieira-Potter VJ, Karamichos D, Lee DJ. Ocular Complications of Diabetes and Therapeutic Approaches. Biomed Res Int. 2016;2016:3801570. doi: 10.1155/2016/3801570. Epub 2016 Mar 28. PMID 27119078
- [Result] El-Agamy A, Alsubaie S. Corneal endothelium and central corneal thickness changes in type 2 diabetes mellitus. Clin Ophthalmol. 2017 Mar 2;11:481-486. doi: 10.2147/OPTH.S126217. eCollection 2017. PMID 28280298
- [Result] Lee JS, Oum BS, Choi HY, Lee JE, Cho BM. Differences in corneal thickness and corneal endothelium related to duration in diabetes. Eye (Lond). 2006 Mar;20(3):315-8. doi: 10.1038/sj.eye.6701868. PMID 15832184
- [Result] Inoue K, Okugawa K, Amano S, Oshika T, Takamura E, Egami F, Umizu G, Aikawa K, Kato S. Blinking and superficial punctate keratopathy in patients with diabetes mellitus. Eye (Lond). 2005 Apr;19(4):418-21. doi: 10.1038/sj.eye.6701497. PMID 15286669
- [Result] Shih KC, Lam KS, Tong L. A systematic review on the impact of diabetes mellitus on the ocular surface. Nutr Diabetes. 2017 Mar 20;7(3):e251. doi: 10.1038/nutd.2017.4. PMID 28319106
- [Result] Murphy PJ, Patel S, Kong N, Ryder RE, Marshall J. Noninvasive assessment of corneal sensitivity in young and elderly diabetic and nondiabetic subjects. Invest Ophthalmol Vis Sci. 2004 Jun;45(6):1737-42. doi: 10.1167/iovs.03-0689. PMID 15161834
- [Result] Dogru M, Katakami C, Inoue M. Tear function and ocular surface changes in noninsulin-dependent diabetes mellitus. Ophthalmology. 2001 Mar;108(3):586-92. doi: 10.1016/s0161-6420(00)00599-6. PMID 11237914
- [Result] Sagdik HM, Ugurbas SH, Can M, Tetikoglu M, Ugurbas E, Ugurbas SC, Alpay A, Ucar F. Tear film osmolarity in patients with diabetes mellitus. Ophthalmic Res. 2013;50(1):1-5. doi: 10.1159/000345770. Epub 2013 Feb 22. PMID 23445780
- [Result] Barbosa FL, Xiao Y, Bian F, Coursey TG, Ko BY, Clevers H, de Paiva CS, Pflugfelder SC. Goblet Cells Contribute to Ocular Surface Immune Tolerance-Implications for Dry Eye Disease. Int J Mol Sci. 2017 May 5;18(5):978. doi: 10.3390/ijms18050978. PMID 28475124
- [Result] Marko CK, Menon BB, Chen G, Whitsett JA, Clevers H, Gipson IK. Spdef null mice lack conjunctival goblet cells and provide a model of dry eye. Am J Pathol. 2013 Jul;183(1):35-48. doi: 10.1016/j.ajpath.2013.03.017. Epub 2013 May 10. PMID 23665202
- [Result] Park Y, Song JS, Choi CY, Yoon KC, Lee HK, Kim HS. A Randomized Multicenter Study Comparing 0.1%, 0.15%, and 0.3% Sodium Hyaluronate with 0.05% Cyclosporine in the Treatment of Dry Eye. J Ocul Pharmacol Ther. 2017 Mar;33(2):66-72. doi: 10.1089/jop.2016.0086. Epub 2016 Dec 8. PMID 27929721
- [Result] Jeon HS, Hyon JY. The Efficacy of Diquafosol Ophthalmic Solution in Non-Sjogren and Sjogren Syndrome Dry Eye Patients Unresponsive to Artificial Tear. J Ocul Pharmacol Ther. 2016 Sep;32(7):463-8. doi: 10.1089/jop.2015.0081. Epub 2016 Jun 13. PMID 27294831
- [Result] Jumblatt JE, Jumblatt MM. Regulation of ocular mucin secretion by P2Y2 nucleotide receptors in rabbit and human conjunctiva. Exp Eye Res. 1998 Sep;67(3):341-6. doi: 10.1006/exer.1998.0520. PMID 9778415
- [Result] Dota A, Sakamoto A, Nagano T, Murakami T, Matsugi T. Effect of Diquafosol Ophthalmic Solution on Airflow-Induced Ocular Surface Disorder in Diabetic Rats. Clin Ophthalmol. 2020 Apr 1;14:1019-1024. doi: 10.2147/OPTH.S242764. eCollection 2020. PMID 32280196
- [Result] Kulkarni AA, Trousdale MD, Stevenson D, Gukasyan HJ, Shiue MH, Kim KJ, Read RW, Lee VH. Nucleotide-induced restoration of conjunctival chloride and fluid secretion in adenovirus type 5-infected pigmented rabbit eyes. J Pharmacol Exp Ther. 2003 Jun;305(3):1206-11. doi: 10.1124/jpet.103.049221. Epub 2003 Mar 20. PMID 12649304
- [Result] Cowlen MS, Zhang VZ, Warnock L, Moyer CF, Peterson WM, Yerxa BR. Localization of ocular P2Y2 receptor gene expression by in situ hybridization. Exp Eye Res. 2003 Jul;77(1):77-84. doi: 10.1016/s0014-4835(03)00068-x. PMID 12823990
- [Result] Tanioka H, Kuriki Y, Sakamoto A, Katsuta O, Kawazu K, Nakamura M. Expression of the P2Y(2) receptor on the rat ocular surface during a 1-year rearing period. Jpn J Ophthalmol. 2014 Nov;58(6):515-21. doi: 10.1007/s10384-014-0342-4. Epub 2014 Sep 2. PMID 25179431
- [Result] Yuko, T.S.; NAKAMURA, M. Stimulatory Effect of Diquafosol Tetrasodium on the Expression of Membrane-Binding Mucin Genes in Cultured Human Corneal Epithelial Cells. Journal of the eye 2011, 28, 425-429.
- [Result] Kaido M, Kawashima M, Shigeno Y, Yamada Y, Tsubota K. Randomized Controlled Study to Investigate the Effect of Topical Diquafosol Tetrasodium on Corneal Sensitivity in Short Tear Break-Up Time Dry Eye. Adv Ther. 2018 May;35(5):697-706. doi: 10.1007/s12325-018-0685-1. Epub 2018 Apr 18. PMID 29671255
- [Result] Ji YW, Kim HM, Ryu SY, Oh JW, Yeo A, Choi CY, Kim MJ, Song JS, Kim HS, Seo KY, Kim KP, Lee HK. Changes in Human Tear Proteome Following Topical Treatment of Dry Eye Disease: Cyclosporine A Versus Diquafosol Tetrasodium. Invest Ophthalmol Vis Sci. 2019 Dec 2;60(15):5035-5044. doi: 10.1167/iovs.19-27872. PMID 31800960
- [Result] Amano S, Inoue K. Effect of topical 3% diquafosol sodium on eyes with dry eye disease and meibomian gland dysfunction. Clin Ophthalmol. 2017 Sep 14;11:1677-1682. doi: 10.2147/OPTH.S148167. eCollection 2017. PMID 29075094
- [Result] Ohashi Y, Munesue M, Shimazaki J, Takamura E, Yokoi N, Watanabe H, Nomura A, Shimada F. Long-Term Safety and Effectiveness of Diquafosol for the Treatment of Dry Eye in a Real-World Setting: A Prospective Observational Study. Adv Ther. 2020 Feb;37(2):707-717. doi: 10.1007/s12325-019-01188-x. Epub 2019 Dec 13. PMID 31834617
- [Derived] Chen J, Zhang Y, Yu S, Zhang Q, He W, Qin G, He X. The Impact of 3% Diquafosol Ophthalmic Solution on Tear Film and Corneal Nerve Density in Patients with Diabetes and Dry Eye Disease: A Randomized Controlled Study. Ophthalmol Ther. 2025 Oct;14(10):2527-2541. doi: 10.1007/s40123-025-01223-x. Epub 2025 Aug 21. PMID 40839332
- [Derived] Chen J, Chen Y, Qin G, Li L, Li M, Cheng Y, Zhuang S, Li Z, Zhang Q, Wu Y, Yang L, Moutari S, Moore JE, Xu L, He W, Yu S, Pazo EE, He X. A protocol for a single center, randomized, controlled trial comparing the clinical efficacy of 3% diquafosol and 0.1% hyaluronic acid in diabetic patients with dry eye disease. Trials. 2023 Dec 12;24(1):803. doi: 10.1186/s13063-023-07818-8. PMID 38087329